CLINICAL TRIAL: NCT04485195
Title: RAFF4 Trial: Vernakalant vs. Procainamide for Acute Atrial Fibrillation in the Emergency Department
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20200402
Record Dates: First submitted 2020-07-14; First posted 2020-07-24 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Atrial Fibrillation
Keywords: Emergency Department; Atrial Fibrillation; Vernakalant; Procainamide
MeSH Terms: conditions — Atrial Fibrillation; Emergencies | interventions — vernakalant; Procainamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vernakalant (Active Comparator): Patients randomized to this arm will receive an initial infusion of 3 mg/kg infused over a 10-minute period by a pre-programmed IV pump.82 For patients ≤ 100 kg the infusion is prepared by adding 25 mL of BRINAVESS 20 mg/mL to 100 mL of diluent creating a total volume of 125 mL at a concentration of 4 mg/mL. For patients > 100 kg the infusion is prepared by adding 30 mL of BRINAVESS 20 mg/mL to 120 mL of diluent creating a total volume of 150 mL at a concentration of 4 mg/mL. For patients weighing ≥ 113 kg, the maximum initial dose is 339 mg (84.7 mL of 4 mg/mL solution).
  Interventions: Drug: Vernakalant
- Procainamide (Active Comparator): Patients randomized to this arm will receive a continuous infusion of IV procainamide with a dose of 15 mg/kg in 500 mL of normal saline given over 60 minutes (maximum dose 1,500 mg), by a pre-programmed pump. While the CAEP Best Practices Checklist suggests an infusion time of 30-60 minutes, we believe that a 60-minute period will avoid some adverse events.
  Interventions: Drug: Procainamide

INTERVENTIONS:
Drug: Vernakalant — an initial infusion of 3 mg/kg infused over a 10-minute period by a pre-programmed IV pump
  Other Names: BRINAVESS
  Arms: Vernakalant
Drug: Procainamide — 15 mg/kg in 500 mL of normal saline given over 60 minutes
  Arms: Procainamide

SUMMARY:
The objective is to compare IV vernakalant to IV procainamide for the ED management of acute AF patients. If vernakalant proves to be more effective, faster, and safer than IV procainamide, this will give clinicians an important alternative for pharmacological cardioversion of acute AF. The investigators propose a pragmatic comparative effectiveness trial entailing an open label, randomized controlled trial at 12 large Canadian EDs. Study subjects will be randomized to 1 of 2 treatment arms: 1) Patients will receive an initial infusion of 3mg/kg of IV vernakalant over 10 minutes, followed by a second dose of 2mg/kg over 10 minutes, if necessary, or 2) Patients will receive a continuous infusion of 15mg/kg of IV procainamide over 60 minutes. The primary aim will be to compare conversion to normal sinus rhythm between the two drugs. The investigators will include stable patients presenting with an episode of acute AF of at least 3 hours duration, where symptoms require urgent management and where immediate cardioversion is a reasonable option. Using the integrated consent model, research assistants will obtain verbal consent from eligible patients.

ELIGIBILITY:
Inclusion Criteria:

The investigators will include stable (see below) patients presenting with an episode of acute non-valvular AF of at least 3 hours duration and no greater than 7 days, where symptoms require urgent management and where immediate cardioversion is a reasonable option because:

1. The patient has been adequately anticoagulated for a minimum of 3 weeks (warfarin and INR > 2.0 or novel oral anticoagulants [dabigatran, rivaroxaban, edoxaban, and apixaban]), or
2. The patient is not adequately anticoagulated for > 3 weeks, has no history of stroke or TIA, and does not have valvular heart disease, AND:

i) onset < 12 hours ago, or ii) if onset 12 - 48 hours ago and there are <2 of these CHADS-65 criteria (age ≥ 65, diabetes, hypertension, heart failure), or iii) negative for thrombus on transesophageal echocardiography. Of note, we will not exclude patients with prior episodes of acute AF. Patients will only be enrolled if the attending physician is confident about time of onset, based upon the patient's symptoms. Physicians are well aware of the importance of this determination and will not attempt to cardiovert patients otherwise.

Exclusion Criteria: The investigators will exclude patients who have any of the reasons listed below.

1. Appropriateness:

   1. unable to understand the study and integrated consent due to language barrier and/or cognitive impairment;
   2. have permanent (chronic) AF;
   3. have valvular heart disease (mitral stenosis, rheumatic or mechanical);
   4. increased risk of stroke because onset not clearly <48 hours and not anticoagulated (or abnormal TEE); or do not meet the inclusion criteria a or b;
   5. deemed unstable and require immediate cardioversion: i) systolic blood pressure <100 mmHg; ii) rapid ventricular preexcitation (Wolff-Parkinson-White syndrome); iii) acute coronary syndrome - chest pain and acute ischemic changes on ECG; or iv) pulmonary edema - severe dyspnea requiring immediate IV diuretic, nitrates, or BIPAP;
   6. primary presentation was for another condition; examples include pneumonia, pulmonary embolism, and sepsis;
   7. convert spontaneously to sinus rhythm prior to randomization;
   8. were previously enrolled in the study; or
   9. have atrial flutter.
2. Safety

   1. has heart failure Class NYHA III or NYHA IV; left ventricular ejection fraction <30%; or has clinical or radiological evidence of acute HF;
   2. has presented with an acute coronary syndrome or acute decompensated heart failure, in the last 30 days; or has had a recent myocardial infarction (< 3 months);
   3. has severe aortic stenosis;
   4. has a systolic blood pressure < 100 mmHg;
   5. has a significantly prolonged QT interval at baseline e.g. uncorrected > 440 msec, congenital or acquired long QT syndrome; or a family history of Long QT syndrome; or ECG shows QTc >460ms (when heart rate >100 measured by the Fridericia formula);
   6. has severe bradycardia (heart rate < 55 bpm), sinus node dysfunction, or second or third degree atrioventricular heart block, in the absence of an in situ properly functioning pacemaker; or, has Brugada syndrome (genetic disease with increased risk of sudden cardiac death);
   7. has received an intravenous antiarrhythmic drug Class I, e.g. procainamide, or Class Ill, e.g. amiodarone or ibutilide, within the prior 4 hours; or currently takes oral class I or III antiarrhythmic drugs other than amiodarone (last dose < 5 half-lives before enrollment);
   8. has received an IV beta-blocker within the 2 hours prior
   9. has hypersensitivity to the active substance or to any of the ingredients of either drug;
   10. has advanced or end-stage liver disease; or
   11. is breast feeding or pregnant (safety not established).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2021-06-17 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2024-11-06 (Actual)

PRIMARY OUTCOMES:
Conversion to sinus rhythm for a minimum duration of 30 minutes | During any time following randomization until 30 minutes past the completion of the drug infusion
  Conversion to and maintenance of sinus rhythm for at least 30 minutes at any time following randomization until 30 minutes past the completion of the drug infusion. Heart rhythm will be determined by an electrocardiogram (ECG).

SECONDARY OUTCOMES:
Normal sinus rhythm | At the time of patient disposition (approximately 3 hours after arrival)
  Being in normal sinus rhythm at the time of ED disposition (discharge or admission). Heart rhythm will be determined by an electrocardiogram (ECG).
Patient disposition (admission or discharge) | At the time of patient admission or discharge (approximately 3 hours after arrival)
  Whether the patient was discharged home or admitted to the hospital.
Length of stay in ED | From time of arrival until time of discharge or admission (approximately 3 hours)
  Length of stay in ED in minutes, from time of arrival to time of discharge or admission
Time to discharge | From time of randomization until time of discharge or admission (approximately 3 hours)
  Time to discharge in minutes, from time of randomization to time of discharge or admission
Time to conversion | From time of infusion start until time of conversion to sinus rhythm (approximately 0 - 90 minutes)
  Time to conversion to sinus rhythm in minutes, from time of start of study drug infusion
Whether the patient required electrical cardioversion | From 30 minutes after the study drug infusion is completed.
  Whether the patient required electrical cardioversion to restore normal sinus rhythm in the ED
Adverse events | 0-12 hours
  will be classified as serious or other, whether occurring 0-2 hours or 2-12 hours after infusion, whether infusion had to be halted or discontinued, or treatment required

OTHER OUTCOMES:
Maintenance of normal sinus rhythm | 30 days post discharge
  Maintenance of normal sinus rhythm at 30 days after ED disposition, to be verified by hospital records, patient report, or by a smartphone application.
Recurrence of acute AF | 30 days
  Recurrence of acute atrial fibrillation requiring an emergency department visit
Death | 30 days
  within 30 days of ED disposition
Stroke | 30 days
  transient ischemic attack, myocardial infarction, or other thromboembolic event within 30 days of ED disposition
Return to normal activities | 30 days
  Return to normal daily activities measured in days

CONTACTS AND LOCATIONS:
Overall Officials: Ian G Stiell, MD, MSc, Principal Investigator — Ottawa Hospital Research Institute
Locations (14):
- Canada (14):
  - University of Alberta Hospital, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Hamilton Health Sciences Centre, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Ottawa Hospital, Ottawa, Ontario
  - St. Michaels, Toronto, Ontario
  - Sunnybrook Hospital, Toronto, Ontario
  - Institut universitaire de cardiologie et de pneumologie de Québec-Université Laval, Laval, Quebec
  - Montreal Heart Institute, Montreal, Quebec
  - Hopital Du Sacre-Coeur, Montreal, Quebec
  - Hopital de L'Enfant-Jesus, Québec, Quebec
  - Hôtel-Dieu de Lévis, Québec, Quebec

REFERENCES:
- [Derived] Stiell IG, Taljaard M, Eagles D, Yadav K, Vadeboncoeur A, Hohl CM, Archambault PM, Birnie D, Brown E, Campbell SG, Chen Y, Clement CM, Cournoyer A, de Wit K, Emond M, Macle L, McRae AD, Mercier E, Morris J, Mohamad G, Nemnom MJ, Nicholls SG, Pare D, Parkash R, Sivilotti M, Thavorn K, Perry JJ. Vernakalant versus procainamide for rapid cardioversion of patients with acute atrial fibrillation (RAFF4): randomised clinical trial. BMJ. 2025 Nov 11;391:e085632. doi: 10.1136/bmj-2025-085632. PMID 41218981